CLINICAL TRIAL: NCT00657371
Title: A Prospective Efficacy Evaluation of the Third Eye Retroscope Auxiliary Imaging System
Brief Title: Efficacy of the Third Eye Retroscope Auxiliary Imaging System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Avantis Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2007-0246
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Results first posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-10

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Colonoscopy; Third Eye Retroscope; Third Eye Retroscope Auxiliary Imaging System; Polypectomy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Third Eye Retroscope (Experimental): Colonoscopy exam using the Third Eye Retroscope device
  Interventions: Device: Third Eye Retroscope Auxiliary Imaging System

INTERVENTIONS:
Device: Third Eye Retroscope Auxiliary Imaging System — A thin, flexible probe that is inserted in a standard colonoscope in order to display very detailed images of the colon tissue.

SUMMARY:
The purpose of this study is to demonstrate efficacy of the Avantis Third Eye Retroscope auxiliary imaging system.

The primary objective of this study is to assess the degree to which incorporating the Third Eye Retroscope auxiliary imaging system in a screening colonoscopy setting results in the detection of additional polyps.

Specifically, the primary goals are to estimate (1) the proportion of polyps detected under this protocol that would have been missed without the Third Eye Retroscope, and (2) the proportion of patients found under this protocol to have polyps who would have incorrectly been classified as polyp-free had the Third Eye Retroscope not been used.

DETAILED DESCRIPTION:
THE STUDY DEVICE:

The Third Eye Retroscope is a thin, flexible probe that can be inserted in a standard colonoscope in order to display very detailed images of the colon tissue. It contains a miniature video camera that allows the doctor to see an additional point of view that looks backward while the regular colonoscope and study device are moved together through the length of the colon.

For you to be eligible to take part in this study, your doctor will check to be sure you have no medical conditions that would increase your risk of having any complications as a result of having the study device used during your colonoscopy.

STUDY PROCEDURES:

If you are found to be eligible to take part in this study, your doctor will perform your colonoscopy exam in the usual manner except that the Third Eye Retroscope device will be used during the exam as well. Your doctor will insert the colonoscope into your rectum in the usual manner and will then insert the study device down a channel inside the colonoscope. You will sign a separate consent form for the colonoscopy, which will describe the procedure and its risks in more detail.

During the exam, you will be awake. If you have chosen to use medications for conscious sedation, you will be drowsy.

FOLLOW-UP PHONE CALL:

About 48 hours (2 days) after the study procedure, you will be called by the research staff to see how you are doing. After this follow-up call, your participation in this study will be over.

This is an investigational study. The Third Eye Retroscope device is commercially available, but it is not FDA approved for this study's purpose. At this time, for this purpose, it is being used in research only. Up to 700 patients will take part in this study. Up to 100 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* The patient is undergoing colonoscopy for screening purposes or for surveillance in follow-up for previous polypectomy.
* The patient is at satisfactory risk for abdominal surgery.
* The patient must understand and provide written consent for the procedure.

Exclusion Criteria:

* Patients who are <50 years or >80 years of age
* Patients who are pregnant.
* Patients with history of colonic resection.
* Patients requiring ongoing anticoagulation therapy.
* Patients with a history of severe cardiovascular, pulmonary, liver or renal disease.
* Patients with hypersensitivity to opioid analgesics.
* Patients with an active systemic infection.
* Patients with suspected chronic stricture potentially precluding complete colonoscopy.
* Patients with major psychiatric disease (dementia, schizophrenia or depression).
* Patients with diverticulitis or toxic megacolon.
* Patients with history of radiation therapy to abdomen or pelvis.
* Patients who are currently enrolled in another clinical investigation in which the intervention might compromise the safety of the patient's participation in this study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2008-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. Bresalier, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (7):
- United States (7):
  - Mayo Clinic, Scottsdale, Arizona
  - El Camino Hospital, Mountain View, California
  - Camino Medical Group Surgi-Center, Sunnyvale, California
  - Indiana University Medical Center, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - U.T.M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Waye JD, Heigh RI, Fleischer DE, Leighton JA, Gurudu S, Aldrich LB, Li J, Ramrakhiani S, Edmundowicz SA, Early DS, Jonnalagadda S, Bresalier RS, Kessler WR, Rex DK. A retrograde-viewing device improves detection of adenomas in the colon: a prospective efficacy evaluation (with videos). Gastrointest Endosc. 2010 Mar;71(3):551-6. doi: 10.1016/j.gie.2009.09.043. Epub 2009 Dec 16. PMID 20018280
- See also: The University of Texas MD Anderson Cancer Center official website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 05, 2008 to May 16, 2010 with recruitment completed in medical settings including university medical centers, ambulatory surgery centers, a community medical center and a physician's office.
Period: Overall Study
Arm/Group | Third Eye Retroscope
Started | 288
Completed | 249
Not Completed | 39
Not completed — Poor bowel preparation | 15
Not completed — Unable to intubate the cecum | 5
Not completed — Protocol Violation | 2
Not completed — Device- related reasons | 13
Not completed — Pre-existing medical condition | 4

BASELINE CHARACTERISTICS:
Population: Of the 288 registered, only 249 had a screening colonoscopy to meet inclusion in the study.
Arm/Group | Third Eye Retroscope
Number analyzed (Participants) | 288
Age Continuous [Mean (Full Range); unit: years] | 63 (6.5) [55 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 156
  Male | 132
Region of Enrollment [Number; unit: participants]
  United States | 288

OUTCOME MEASURES:

1. Primary Outcome: Increase (Percent) of Polyps Detected That Would Have Been Missed Without the Third Eye Retroscope (TER)
Description: After cecal intubation, the disposable TER was inserted through the instrument channel of the colonoscope. During withdrawal, the forward and retrograde video images were observed simultaneously on a wide-screen monitor. A 2 year study period was used to collect colonoscopy exam results.
Time Frame: Total 30 minutes procedure time with TER use.
Measure: Number; unit: percent of polyps
Units Other Than Participants: Polyps
Arm/Group | Third Eye Retroscope
Number analyzed (Participants) | 249
Number analyzed (Polyps) | 257
percent of polyps | 13.2

2. Secondary Outcome: Number Participants With Polyps Who Would Have Incorrectly Been Classified as Polyp-free Had the Third Eye Retroscope Not Been Used.
Description: Colonoscope and TER use where during TER withdrawal forward and retrograde video images observed simultaneously on a wide-screen monitor for purpose of detecting polyps. Colonoscopy procedures completed in approximately 30 minutes total.
Time Frame: 2 year study period to collect colonoscopy exam results
Reporting Status: Not Posted

3. Primary Outcome: Number Polyps Detected With the Standard Colonoscope and Third Eye Retroscope (TER)
Description: as for outcome 1
Time Frame: Total 30 minutes procedure time with TER use.
Population: Those polyps reported for Third Eye Retroscope were additional, located behind folds and then found with the colonscope only because they were first detected with the Third Eye Retroscope.
Measure: Number; unit: polyps
Units Other Than Participants: Polyps
Arm/Group | Third Eye Retroscope
Number analyzed (Participants) | 249
Number analyzed (Polyps) | 257
polyps
  Standard Colonoscope (Total) | 257
  Third Eye Retroscope | 34

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Third Eye Retroscope
Serious Adverse Events (participants affected / at risk) | 0/288
Other Adverse Events (participants affected / at risk) | 0/288

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No